CLINICAL TRIAL: NCT06320626
Title: Pharmacokinetic-guided Dosing of Emicizumab in Congenital Haemophilia A Patients - The DosEmi Study
Brief Title: Pharmacokinetic-guided Dosing of Emicizumab
Acronym: DosEmi
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Kathelijn Fischer (Other)
Collaborators: Erasmus Medical Center (Other); Amsterdam University Medical Center (Other); Leiden University Medical Center (Other); Radboud University Medical Center (Other); Maastricht University Medical Center (Other); University Medical Center Groningen (Other); HagaZiekenhuis (Other); Dutch Society of Haemophilia Patients (Unknown)
Responsible Party: Sponsor-Investigator, Kathelijn Fischer, Principal Investigator, UMC Utrecht
Organization: UMC Utrecht (Other)
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 22-571
Record Dates: First submitted 2024-02-28; First posted 2024-03-20 (Actual); Last update posted 2024-03-20 (Actual); Status verified 2024-03

CONDITIONS: Hemophilia A With Inhibitor; Hemophilia A Without Inhibitor; Hemophilia A, Severe; Adolescent; Child; Adult
Keywords: Emicizumab; Hemophilia A; Monoclonal antibodies; PK-guided dosing; Hemorrhage
MeSH Terms: conditions — Hemophilia A; Hemorrhage | interventions — emicizumab

STUDY DESIGN:
Intervention Model Description: * PK-guided dosing - Intervention group (12M): Subjects with emicizumab concentration of ≥ 40 μg/mL will receive individualized PK-guided dose reduction of emicizumab targeted at a Ctrough of 30μg/mL. The validated population PK model is based on published population PK and PK/PD modelling studies. (9,10,15)
  * PK-Guided dosing - Non-intervention group (12M): Subjects with emicizumab concentration of 25-39 μg/mL will continue on their current dose regimen and will be followed according to the same assessment schedule as the Intervention Group. Only subjects with emicizumab plasma concentration < 25 μg/mL will be adjusted in dosing regimen according to local protocol. These subjects will be followed for selective safety data only.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Conventional dosing - open label (Other): Patients will be followed 6 months retrospectively and 6 months prospectively on conventional dosing.
  Interventions: Other: Emicizumab - PK-guided dose reduction; Other: Emicizumab - Dosis continuation group; Other: Emicizumab - Dose adjustment group
- PK-guided dosing - open label (Other): Patients with emicizumab concentration of ≥ 40 μg/mL will receive individualized PK-guided dose reduction of emicizumab targeted at a Ctrough of 30μg/mL. Patients will be followed for 12 months on reduced dosing.
  Interventions: Other: Emicizumab - PK-guided dose reduction
- No intervention continuation - open label (Other): Patients with emicizumab concentration of 25-39 μg/mL will continue on their current dose regimen. Patients will be followed for 12 months on current dosing.
  Interventions: Other: Emicizumab - Dosis continuation group
- No intervention adjusted - open label (Other): Patients with emicizumab plasma concentration < 25 μg/mL will be adjusted in dosing regimen according to local protocol. Patients will be followed for selective safety data only.
  Interventions: Other: Emicizumab - Dose adjustment group

INTERVENTIONS:
Other: Emicizumab - PK-guided dose reduction — PK-guided dose reduction emicizumab targeted at a Ctrough of 30μg/mL.
  Other Names: Hemlibra
  Arms: Conventional dosing - open label; PK-guided dosing - open label
Other: Emicizumab - Dosis continuation group — Continue on their current dose regimen
  Other Names: Hemlibra
  Arms: Conventional dosing - open label; No intervention continuation - open label
Other: Emicizumab - Dose adjustment group — Adjusted in dosing regimen according to local protocol
  Other Names: Hemlibra
  Arms: Conventional dosing - open label; No intervention adjusted - open label

SUMMARY:
The goal of this multicentre, prospective, open-label, cross-over clinical study is to determine whether individualized PK-guided dosing of emicizumab is non-inferior to conventional dosing of emicizumab in the prevention of bleeding in congenital haemophilia A patients.

DETAILED DESCRIPTION:
Haemophilia A is an X-linked hereditary bleeding disorder resulting from a deficiency or dysfunction of endogenous coagulation factor VIII (FVIII). Persons with haemophilia A (PwHA) suffer from spontaneous or provoked bleeding, predominantly into major joints, which eventually lead to painful and chronic disabling arthropathy. The primary goal in clinical management of haemophilia A is prevention of bleeding by self-administration of FVIII concentrates via intravenous injections.

Prophylaxis with FVIII concentrates has effectively reduced treated bleeds from an annual average of 20-30 to 1-4. However, in approximately 30% of PwHA anti-FVIII antibodies (known as inhibitors) develop that interfere with FVIII replacement therapy. PwHA who develop inhibitors require alternative suboptimal therapy with (costly) bypassing agents (BPA).

The first approved non-factor therapy is the bispecific, FVIII-mimicking antibody, emicizumab (Hemlibra®), which came available in the Netherlands in July 2018. Emicizumab is a humanized, bispecific antibody connecting factor IX and factor X enabling the activation of FX and subsequent thrombin generation. Emicizumab has shown to be highly effective prophylaxis in PwHA by achieving a complete eradication of treated bleeds in around 80% of PwHA (n = 374) during the second 24-week interval of treatment. Furter advantages of emicizumab are the subcutaneous administration and less frequent dosing intervals every 1, 2 or 4 weeks due to a long half-life (t ½: 28 days). Despite many PwHA are candidate for prophylaxis with emicizumab, cost limit widespread access.

Currently, emicizumab is approved by F. Hoffmann-La Roche® with a loading dose of 3 mg/kg/week for four weeks and a maintenance dose of 1.5 mg/kg/week, 3 mg/kg/2 weeks or 6 mg/kg/4 weeks. These dose regimens were based on a pharmacometric approach instead of a dose finding study, and targeted a trough concentration (Ctrough) of 45 µg/ml by using pharmacokinetic (PK)simulations. Meanwhile long-term bleed data from the phase III and IV studies by the pharmaceutical company were included in pharmacokinetic (PK) and pharmacodynamic (PD) modelling studies, and the effective Ctrough was suggested at 30 µg/ml.

Although this Ctrough of 30 µg/ml is substantially lower than the previous Ctrough (45 µg/ml), the dose regimens were not adjusted. Conventional dosing leads to mean concentrations of 55 µg/ml with two thirds of the observations between 40 and 70 µg/ml (i.e., SD of ±15 µg/ml). Emicizumab has been approved based on fixed body-weight-based dosing and therefore the concentration target might have been kept higher to avoid lower effectivity due to inter-patient variability. However, reduced dosing of emicizumab, either by extending the dosing interval or lowering the dose, without sacrificing its efficacy has been reported in small case series.

Therefore, the investigators hypothesized that lower dosing of emicizumab targeted at Ctrough 30 μg/mL, is equally as effective and less costly in preventing bleeds as conventional dosing of emicizumab, and designed the DosEmi study to investigate the hypothesis in a large prospective cohort of adult and paediatric PwHA.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of congenital haemophilia A, with a baseline endogenous FVIII of <6 IU/ml
* Aged > 1 year at inclusion (inclusion of children 1-16 years after favourable interim-analysis see protocol)
* Receiving conventional dosing of emicizumab (6 mg/kg/4 weeks with varying intervals) for a duration of at least 12 months prior to inclusion;
* Having good bleeding control, defined as:

i No spontaneous joint/muscle bleeds in the previous 6 months AND ii A maximum of two treated (traumatic) bleeds in the previous 6 months.

* Willing and able to provide written informed consent, either by the subject or its parents/legal guardian
* Willing to provide bleeding assessment information
* Willing to adhere to the medication regimen

Exclusion Criteria:

* Acquired haemophilia A

Min Age: 1 Year | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Gender Based: Yes
Enrollment: 95 (Estimated)
Dates: Start 2022-09-08 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients without treated bleeds | 12 months
  Comparison proportion treated bleeds 6 months before (conventional) and after intervention (PK-guided dosing)

SECONDARY OUTCOMES:
Proportion of patients without treated bleeds | 24 months
  Comparison proportion without treated bleeds 12 months before (conventional) and after intervention (PK-guided dosing)
Proportion of patients without spontaneous joint- or muscle bleeds | 24 months
  Comparison proportion without spontaneous joint- or muscle bleeds 6 and 12 months before and after intervention.
Annualized bleeding rate (ABR) of treated bleeds, including joint bleeds and sport-induced bleeds | 24 months
  Comparison annualized bleeding rate 6 and 12 months before and after intervention.
To compare cost-effectiveness between conventional dosing and individualized PK-guided dosing of emicizumab | 24 months
  Direct and indirect medical costs: Direct medical costs are predominantly determined by consumption of emicizumab, additional FVIII, and/or bypassing agents, extracted from the hospital's pharmacy records. These data are highly reliable, as this medication is exclusively distributed by haemophilia treatment centers. Indirect medical costs: are number of (emergency) hospital visits, bleeding related hospital admissions and/or unscheduled surgeries, and days lost from work/school (for patients and/or caregivers).
To assess the cumulative number of coagulation factor (sc. and/or iv.) of per year. | 24 months
  Assessment of the cumulative number of sc. and/or iv. Injections related to coagulation correction.
To assess the performance of the population PK model | 12 months
  Predictive performance of the MAP Bayesian procedure used for the dose adaptation procedure, defined as % of patients within ±20% of target level/within the target level of 25-39 µg/mL of emicizumab.
To investigate whether direct joint health remains stable measured by physical examination when switching to lower-dosed emicizumab compared to conventional treatment | 12 months
  Joint status will be measured by physical examination (Haemophilia Joint Health Score; HJHS),
To investigate whether direct joint health remains stable measured by ultrasound when switching to lower-dosed emicizumab compared to conventional treatment | 12 months
  Joint status will be measured by ultrasound (if available, according to the HEAD US score).
To investigate if indirect joint health, as measured by biomarkers, remains stable when switching to lower doses of emicizumab compared to conventional treatment. | 12 months
  biomarker assessment for inflammation and joint and cartilage turnover in blood. The biomarkers comprising origin of different joint tissues will be selected and adopted based on the literature on osteoarthritis, which is a rapidly changing area of research.
To investigate if indirect joint health, as measured by biomarkers, remains stable when switching to lower doses of emicizumab compared to conventional treatment. | 12 months
  biomarker assessment for inflammation and joint and cartilage turnover in urine.The biomarkers comprising origin of different joint tissues will be selected and adopted based on the literature on osteoarthritis, which is a rapidly changing area of research.
To investigate whether Health Related Quality of Life (HR-QoL) are similar in patients receiving conventional dosing compared with PK-guided dosing of emicizumab. | 12 months
  Health related quality of life will be assessed with EuroQol Five Dimensions Health Questionnaire (Youth) EQ5D(Y).
To investigate whether Health Related Quality of Life (HR-QoL) are similar in patients receiving conventional dosing compared with PK-guided dosing of emicizumab. | 12 months
  Health related quality of life will be assed with PROMIS instruments (Physical Function/mobility and Pain Interference short forms).
To investigate whether sports participation are similar in patients receiving conventional dosing compared with PK-guided dosing of emicizumab. | 12 months
  Sports participation (type, duration, frequency) will be assessed with Modifiable Activities Questionnaire (MAQ).
To investigate whether thrombin generation parameters can be used as a pharmacodynamic (PD) biomarker for emicizumab treatment efficacy. | 12 months
  To measure coagulation potential, blood samples will be collected to measure thrombin generation (Peak Height and ETP)
To assess and monitor pain during emicizumab administration | 12 months
  Assessment of pain during emicizumab administration by Visual Analogue Scale (scale 0-10)

CONTACTS AND LOCATIONS:
Overall Officials: Study Officials Fischer, Dr, MD, Principal Investigator — UMC Utrecht
Locations (8):
- Netherlands (8):
  - Radboud University Medical Center, Nijmegen, Gelderland
  - Maastricht University Medical Center, Maastricht, Limburg
  - Amsterdam University Medical Center, Amsterdam, North Holland
  - Leids Universitair Medisch Centrum, Leiden, South Holland
  - Erasmus University Medical Center, Rotterdam, South Holland
  - HagaZiekenhuis, The Hague, South Holland
  - University Medical Center Groningen, Groningen
  - University Medical Center Utrecht, Utrecht

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP
URL: http://bmjopen.bmj.com/content/13/6/e072363.long

REFERENCES:
- [Background] Donners A, van der Zwet K, Egberts ACG, Fijnvandraat K, Mathot R, Kruis I, Cnossen MH, Schutgens R, Urbanus RT, Fischer K. DosEmi study protocol: a phase IV, multicentre, open-label, crossover study to evaluate non-inferiority of pharmacokinetic-guided reduced dosing compared with conventional dosing of emicizumab in people with haemophilia A. BMJ Open. 2023 Jun 26;13(6):e072363. doi: 10.1136/bmjopen-2023-072363. PMID 37369395
- [Background] Berntorp E, Fischer K, Hart DP, Mancuso ME, Stephensen D, Shapiro AD, Blanchette V. Haemophilia. Nat Rev Dis Primers. 2021 Jun 24;7(1):45. doi: 10.1038/s41572-021-00278-x. PMID 34168126
- [Background] Blanchette VS, Key NS, Ljung LR, Manco-Johnson MJ, van den Berg HM, Srivastava A; Subcommittee on Factor VIII, Factor IX and Rare Coagulation Disorders of the Scientific and Standardization Committee of the International Society on Thrombosis and Hemostasis. Definitions in hemophilia: communication from the SSC of the ISTH. J Thromb Haemost. 2014 Nov;12(11):1935-9. doi: 10.1111/jth.12672. Epub 2014 Sep 3. No abstract available. PMID 25059285
- [Background] Srivastava A, Santagostino E, Dougall A, Kitchen S, Sutherland M, Pipe SW, Carcao M, Mahlangu J, Ragni MV, Windyga J, Llinas A, Goddard NJ, Mohan R, Poonnoose PM, Feldman BM, Lewis SZ, van den Berg HM, Pierce GF; WFH Guidelines for the Management of Hemophilia panelists and co-authors. WFH Guidelines for the Management of Hemophilia, 3rd edition. Haemophilia. 2020 Aug;26 Suppl 6:1-158. doi: 10.1111/hae.14046. Epub 2020 Aug 3. No abstract available. PMID 32744769
- [Background] Callaghan MU, Negrier C, Paz-Priel I, Chang T, Chebon S, Lehle M, Mahlangu J, Young G, Kruse-Jarres R, Mancuso ME, Niggli M, Howard M, Bienz NS, Shima M, Jimenez-Yuste V, Schmitt C, Asikanius E, Levy GG, Pipe SW, Oldenburg J. Long-term outcomes with emicizumab prophylaxis for hemophilia A with or without FVIII inhibitors from the HAVEN 1-4 studies. Blood. 2021 Apr 22;137(16):2231-2242. doi: 10.1182/blood.2020009217. PMID 33512413
- [Background] Yoneyama K, Schmitt C, Kotani N, Levy GG, Kasai R, Iida S, Shima M, Kawanishi T. A Pharmacometric Approach to Substitute for a Conventional Dose-Finding Study in Rare Diseases: Example of Phase III Dose Selection for Emicizumab in Hemophilia A. Clin Pharmacokinet. 2018 Sep;57(9):1123-1134. doi: 10.1007/s40262-017-0616-3. PMID 29214439
- [Background] Retout S, Schmitt C, Petry C, Mercier F, Frey N. Population Pharmacokinetic Analysis and Exploratory Exposure-Bleeding Rate Relationship of Emicizumab in Adult and Pediatric Persons with Hemophilia A. Clin Pharmacokinet. 2020 Dec;59(12):1611-1625. doi: 10.1007/s40262-020-00904-z. PMID 32504271
- [Background] Jonsson F, Schmitt C, Petry C, Mercier F, Frey N, Retout S. Exposure-Bleeding Count Modeling of Emicizumab for the Prophylaxis of Bleeding in Persons with Hemophilia A with/Without Inhibitors Against Factor VIII. Clin Pharmacokinet. 2021 Jul;60(7):931-941. doi: 10.1007/s40262-021-01006-0. Epub 2021 Mar 12. PMID 33709296
- [Background] Donners AAMT, Rademaker CMA, Bevers LAH, Huitema ADR, Schutgens REG, Egberts TCG, Fischer K. Pharmacokinetics and Associated Efficacy of Emicizumab in Humans: A Systematic Review. Clin Pharmacokinet. 2021 Nov;60(11):1395-1406. doi: 10.1007/s40262-021-01042-w. Epub 2021 Aug 13. PMID 34389928
- [Background] Lehtinen AE, Lassila R. Do we need all that emicizumab? Haemophilia. 2022 Mar;28(2):e53-e55. doi: 10.1111/hae.14483. Epub 2021 Dec 30. No abstract available. PMID 34970820
- [Background] Chuansumrit A, Sirachainan N, Jaovisidha S, Jiravichitchai T, Kadegasem P, Kempka K, Panuwannakorn M, Rotchanapanya W, Nuntiyakul T. Effectiveness of monthly low dose emicizumab prophylaxis without 4-week loading doses among patients with haemophilia A with and without inhibitors: A case series report. Haemophilia. 2023 Jan;29(1):382-385. doi: 10.1111/hae.14707. Epub 2022 Nov 29. No abstract available. PMID 36446746
- [Background] Bansal S, Donners AAMT, Fischer K, Kshirsagar S, Rangarajan S, Phadke V, Mhatre S, Sontate B, Silva M, Ansari S, Shetty S. Low dose emicizumab prophylaxis in haemophilia a patients: A pilot study from India. Haemophilia. 2023 May;29(3):931-934. doi: 10.1111/hae.14785. Epub 2023 Apr 8. No abstract available. PMID 37029771
- Available data/document: Study Protocol: 37369395 — http://bmjopen.bmj.com/content/13/6/e072363.long — Published study protocol